CLINICAL TRIAL: NCT06026631
Title: Lipidomic Characterization in Non-metastatic Breast Cancer Women Undergoing Surgery: a Pilot Study.
Acronym: BreCaLip
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Magno Stefano, Head of UOS Breast Integrative Oncology, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FPGemelliIRCCS4663
Record Dates: First submitted 2023-08-10; First posted 2023-09-07 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Lipid Cell; Tumor; Nutrition Related Cancer; Body Weight
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (breast cancer) (Experimental): Lipidomic analysis for breast cancer patients
  Interventions: Procedure: Lipidomic analysis for breast cancer patients
- Control arm (healthy subject) (Other): Lipidomic analysis for healthy subjects
  Interventions: Procedure: Lipidomic analysis for breast cancer patients

INTERVENTIONS:
Procedure: Lipidomic analysis for breast cancer patients — Lipidomic analysis for breast cancer patients

SUMMARY:
The goal of this clinical trial is to learn about breast cancer lipodome signature in patients waiting for surgery with different Body Mass Index.

The main question it aims to answer are:

* To highlight a specific lipidome molecular signature for breast cancer patients overweight and obese (BMI > 25 Kg/m2) compared with patients of normal weight (BMI<25 kg/m2).
* Evaluate the effect of the pool of biochemical, nutritional and anatomical-pathological data of breast cancer patients and the correlation between molecular profile and body weight.

ELIGIBILITY:
Patients

* Age <65 years (not to have influence on functioning of desaturase enzymes that decline with older ages).
* Neoplastic pathology: primary invasive breast cancer or ductal in situ (DCIS) newly diagnosed, in the pre-operative phase and which has not already undergone chemo- or radiotherapy.
* Absence of serious intestinal and hepatic pathologies, diabetes, both insulin-dependent and in hypoglycaemic treatment or other pancreatic affection, thyroid affections in pharmacological treatment.
* Absence of supplementation with omega-3 based supplements for at least 6 months.
* Homogeneous distribution by BMI (1:1 ratio subjects with BMI≥25 and BMI<25, respectively).
* Informed consent to participate in the study.

controls

* Age <65 years;
* Not be affected by cancer;
* BMI <25kg/m2;
* Informed consent to participate in the study

Exclusion Criteria:

patients

* Age ≥65 years (would affect the functioning of desaturase enzymes that decline with older age).
* Invasive primary breast cancer or ductal in situ (DCIS) previously treated with chemo- or radiotherapy.
* Metastasis at diagnosis.
* Presence of serious intestinal and hepatic pathologies.
* Presence of diabetes, both insulin-dependent and in hypoglycaemic treatment or other pancreatic disease, thyroid disease in pharmacological treatment.
* Supplementation with omega-3 based supplements for at least 6 months.
* Failure to sign the informed consent to participate in the study.

controls

* Age ≥65 years;
* Suffering from tumor pathology;
* BMI ≥25kg/m2;
* Refusal to sign informed consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Correlation lipidome and BMI | First day
  Evaluate the correlation between some biomarkers derived from the lipidomic study (e.g. palmitic acid, stearic acid, oleic acid, palmitoleic acid and sapienic acid, arachidonic acid, dihomogammalinolenic acid, EPA, DHA, etc…) according to the BMI class considered.

SECONDARY OUTCOMES:
Correlation lipidome and nutrition/anatomical-pathological | First day
  Evaluate the correlation of molecular data with biochemical, nutritional and anatomical-pathological data of the patients and of the tumor (NLR -neutrophil-to-lymphocyte ratio), glycemia, cholesterol, blood pressure, triglycerides; TILs (percentage of lymphocytic infiltrate) and Ki67 (proliferation factor) on the surgical sample; W/H ratio, % FAT, % LEAN, phase angle at bioimpedance analysis in the study sample.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Magno, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No